CLINICAL TRIAL: NCT06351540
Title: Examining the Role of Tolerance on Dose-dependent Effects of Acute THC on Oculomotor and Cognitive Performance
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00332797; R21DA056687 (NIH)
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cannabis Use; Impaired Driving; Cognitive Impairment
Keywords: cannabis; THC; impairment
MeSH Terms: conditions — Cognitive Dysfunction; Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: double-blind, placebo-controlled, within-subjects crossover design
Who Masked: Participant, Investigator
Masking Description: placebo controlled, double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0 mg THC (Placebo Comparator): Inhaled Cannabis - 0 mg THC
  Interventions: Drug: Cannabis
- 5 mg THC (Experimental): Inhaled cannabis - 5 mg THC
  Interventions: Drug: Cannabis
- 30 mg THC (Experimental): Inhaled cannabis - 30 mg THC
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Cannabis — cannabis with 0, 5, or 30 mg THC will be inhaled via vaporization

SUMMARY:
The purpose of this research is to determine the extent to which oculomotor function accurately detects THC-impairment, if cannabis use experience impacts this detection threshold, and to examine how the oculomotor index corresponds to a measure of sustained attention. A double-blind, placebo-controlled, within-subjects crossover design will be used to examine the dose-effects of THC (0, 5mg, 30mg) on oculomotor performance tasks and a sustained attention task in frequent and infrequent cannabis users. Results from the study will advance the investigators' understanding of the effect of THC and cannabis use frequency on oculomotor function and sustained attention, and will directly inform the validity of the investigators' oculomotor platform for identifying acute THC- induced impairment in frequent and infrequent users.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: Healthy non-treatment seeking adults (age 18 to 60, N = 40) who report
* (a) infrequent cannabis use defined as at least one reported use in the past year with a negative THC urine toxicology at baseline, or
* (b) report frequent cannabis use defined as > 5 days per week for > 1 year with a positive THC urine toxicology at baseline.

These criteria were selected to target individuals with low and high-frequency cannabis use in order to examine the direct effect of tolerance on study outcome measures.

Exclusion Criteria:

* (1) meet DSM-V criteria for substance use disorders other than tobacco, cannabis, or caffeine,
* (2) are currently receiving or interested in immediately receiving behavioral treatment or medication for cannabis cessation,
* (3) current use of any medications that could affect study outcomes,
* (4) test positive for drugs of abuse (other than cannabis) and/or breath alcohol test at study admission,
* (5) have a current physical or mental illness judged by the study team to negatively impact participant safety or scientific integrity,
* (6) are currently pregnant, planning to become pregnant in the next three months or are currently breastfeeding,
* (7) have a history of clinically significant cardiac arrhythmias or vasospastic disease (e.g. Prinzmetal's angina), or (8) are currently enrolled in another clinical trial or have received any drug as part of a research study within 30 days of study participation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Commission Errors | pre-administration, post-administration, 2, 4 hours
  The Conners Continuous Performance Test (CPT) will be used to assess sustained attention. Commission errors is measured by calculating the number of trials participants incorrectly push the spacebar in the presence of "X" stimulus.
Omission Errors | pre-administration, post-administration, 2, 4 hours
  The Conners Continuous Performance Test (CPT) will be used to assess sustained attention. Omission errors is measured by calculating the number of trials participants fail to push the spacebar in the presence of a letter that is not an "X" stimulus.
Reaction Time | pre-administration, post-administration, 2, 4 hours
  The Conners Continuous Performance Test (CPT) will be used to assess sustained attention. Reaction time is measured by calculating the duration between the presentation of a letter other than "X", and the correct response of a spacebar push.
Reaction Time Standard Error | pre-administration, post-administration, 2, 4 hours
  The Conners Continuous Performance Test (CPT) will be used to assess sustained attention. Reaction time standard error is measured by calculating the standard error of the mean of the reaction time.
Visuomotor Index | pre-administration, post-administration, 2, 4 hours
  The visuomotor index score is calculated by mathematically integrating five measures of oculomotor fixation performance and two measures of accuracy into a single score during fixation and accuracy tasks, respectively. Test of visual fixation to measure microsaccades, spontaneous nystagmus, and gaze-evoked nystagmus.

SECONDARY OUTCOMES:
Saccade Speed | Pre-administration, post-administration, 2, 4 hours
  Measures how quickly participants look back and forth between two spots as possible during the oculomotor task.
Visually Guided Oculomotor Performance | Pre-administration, post-administration, 2, 4 hours
  Measures how quickly and accurately participants move their eyes to a cue as soon as it appears on the oculomotor task.
Antisaccade | Pre-administration, post-administration, 2, 4 hours
  Measures voluntary eye movement in the direction opposite to the side in which a visual cue is presented.
Memory-Guided | Pre-administration, post-administration, 2, 4 hours
  Measures how quickly gaze is shifted directly and accurately to a remembered cue position.

CONTACTS AND LOCATIONS:
Overall Officials: Dustin C Lee, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No